CLINICAL TRIAL: NCT03379207
Title: Innate Immunity During Community Acquired Pneumonia: A Translational Approach
Brief Title: Innate Immune Response During Community Acquired Pneumonia
Acronym: ImPACT
Status: Terminated | Type: Observational
Why Stopped: A new project has been started. It extends ImPACT, with more financial resources and with scientific questions that have evolved.
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHAO17/YJ-ImPACT
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Community-acquired Pneumonia; Acute Respiratory Distress Syndrome; Innate Immunity
Keywords: Community-acquired Pneumonia; Acute Respiratory Distress Syndrome; Innate Immunity; Non Conventional T Lymphocytes
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for all participants; Tracheal aspirations for invasively ventilated patients; Broncho alveolar lavage fluid when available (indication left at the discretion of the investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "Community Acquired Pneumonia" group: Participants admitted to Intensive Care Unit (ICU) of University Hospital of Tours (France) for Community Acquired Pneumonia.
  Interventions:
  * Blood samples for research purpose, taken whenever possible during blood sampling for routine purpose, at inclusion, day 1, 7, and every week during ICU stay Tracheal Aspirates for research purpose: only for mechanically ventilated participants, at inclusion, day 1, 7, and and every week during ICU stay
  * Surplus of Broncho-alveolar lavage fluid: only if performed for diagnosis purpose by the treating investigator (indication left at his discretion)
  Interventions: Other: Blood samples; Other: Tracheal Aspirates; Other: Surplus of Broncho-alveolar lavage fluid
- "Control" group: Participants admitted to Intensive Care Unit of University Hospital of Tours (France) for whom invasive mechanical ventilation is required for an estimated duration of at least 48h, without diagnosis of pneumonia or shock.
  Interventions:
  * Blood samples for research purpose, taken whenever possible during blood sampling for routine purpose, at inclusion, day 3, 8, and 15 during ICU stay Tracheal Aspirates for research purpose: at inclusion, day 3, 8, and 15 during invasive mechanical ventilation period,
  * Surplus of Broncho-alveolar lavage fluid: only if performed for diagnosis purpose by the treating investigator (indication left at his discretion)
  Interventions: Other: Blood samples; Other: Tracheal Aspirates; Other: Surplus of Broncho-alveolar lavage fluid

INTERVENTIONS:
Other: Blood samples — Blood samples for research purpose, taken whenever possible during blood sampling for routine purpose
Other: Tracheal Aspirates — Only for mechanically ventilated participants.
Other: Surplus of Broncho-alveolar lavage fluid — Only if performed for diagnosis purpose by the treating investigator : indication left at his discretion

SUMMARY:
Community acquired pneumonia (CAP) is a major cause of morbidity and mortality worldwide. Despite recent improvement in acute management (specifically for administration of antibiotics) many severe presentations of pneumonia worsen, progressing to Acute Respiratory Distress Syndrome (ARDS), a clinical entity with 40% hospital mortality.

Dysregulation of immune response is thought to be largely implicated in severe pneumonia progressing to ARDS. Notably, experimental studies have recently suggested the implication of non-conventional T lymphocytes and innate cells in this immunopathology. However, no data are available in Humans in clinical settings.

This study aims to explore the role of non-conventional T cells in pneumonia and ARDS, in participants. For this purpose, 100 participants admitted to Intensive Care Unit (ICU) with a diagnosis of CAP will be included, and 50 "control" participants with no pneumonia nor shock. Presence and functionality of non-conventional T cells and innate cells will be explored using flow-cytometry and ex-vivo stimulation, alongside with cytokines productions. These analyses are conducted in the blood, and, for invasively ventilated participants, in tracheal aspirates or broncho-alveolar fluids if available. For each participants included, the analyses are conducted at different time-points during ICU stay: inclusion, day 3, day 8 and day 15. Moreover, participants with ARDS, for whom a post-ICU follow-up program is normally established after discharge, will have blood analysis from blood samples taken during the follow-up visit up to 8 months after inclusion.

Immunophenotypage and functionality of non-conventional T cells and innate cells will be compared to clinical parameters and their evolution, between "CAP" participants and "Control" participants", and for each participants, according to the different time-point of analysis, in order to better understand dynamic of innate immunity during pneumonia and ARDS.

DETAILED DESCRIPTION:
- Clinical and scientific background:

Community acquired pneumonia is a major cause of morbidity and mortality worldwide. Despite recent improvement in acute management (specifically for administration of antibiotics), severe pneumonia can worsen and ultimately progressing to Acute Respiratory Distress Syndrome (ARDS), a clinical entity with an inacceptable 40% hospital mortality. From a pathophysiological point of view, ARDS is characterized by a deregulation of pulmonary inflammation initially triggered by the local aggression, which is, in two-third of the cases, a pneumonia. Alteration of tissue repair is another major characteristic of this entity. So far, the scientific knowledge on this pathophysiology did not translate into specific therapy that could modulate efficiently the inflammatory response and to control the progression from pneumonia to ARDS, and/or to improve tissue repair. Thus, a complete reconsideration of the pathophysiological mechanisms is mandatory. Recent progresses in mucosal biology and innate immunity give interesting new opportunities. Specifically, recently discovered unconventional T cells have shown to be major actors in shaping and modulating early immune responses in the lung mucosa during microbial aggressions and for secondary tissue repair. However, these evidences are limited to pre-clinical models. In many other human diseases (oncology, immune diseases), these sub-populations are already being explored as potential targets for immune therapies.

- Objective of the study:

The aim of this study is to explore potential implications of unconventional T cells during human severe pneumonia and ARDS.

This translational study will complement experimental approaches currently undertaken in the laboratory exploring the role of unconventional T cells in murine models of severe pneumonia and ARDS.

- Design:

This is a prospective single-center study including participants admitted in Intensive Care Department of the university hospital of Tours for community-acquired pneumonia. Given the exploratory nature of the study, we designed a "control" group of participants admitted to ICU without evident signs of pneumonia and shock.

Number of participants: 300 for "pneumonia" group, and 50 for "control" group

- Interventions and analysis:

Blood samples will be collected at inclusion, day 3, 8 and 15 during patient's stay in ICU. For mechanically ventilated participants, tracheal aspirates will be also collected at the same timing. If available, broncho-alveolar lavages will be also collected. If ARDS or Ventilator Associated Pneumonia (VAP) are subsequently diagnosed, supplemental blood and tracheal aspirates samples will be collected.

Blood samples and airway fluid samples will be treated to perform flow cytometry analysis for immunophenotypage (cellular content). In some cases, intra-cellular staining will be performed to assess cytokine production and/or transcription factor expression. Functions of unconventional T cells will also be performed after ex vivo stimulation on purified population (cell sorting). Cytokine level sand transcriptomic analyses will also be performed on blood samples.

Clinical characteristics (including respiratory parameters, blood gas, organ dysfunctions, survival at day 28 and day 90) will also be collected. Thus, frequency, activation status and functions of unconventional T cells will be dynamically analyzed in regard of clinical evolution within-individuals and across pneumonia vs control groups. A particular focus will be made on respiratory parameters (ventilation mode, and for participants with ARDS, P/F ratio, driving pressure), organ dysfunctions (as measured by SOFA score), and microbial documentation of the pneumonia.

Moreover, participants treated for ARDS are usually followed in a post-ICU follow-up clinic program in the ICU where the research is conducted. Thus, investigators will perform analysis of the unconventional T cell compartment (blood samples) in the participants firstly enrolled in the study. This will allow exploration of long-term imprinting on the innate immune response after the initial trigger.

ELIGIBILITY:
Inclusion criteria:

"Pneumonia" group:

* Admission to the Intensive Care Units or Pneumonia service of Tours University Hospital or Intensive Care Unit or Limoges University Hospital
* Initial diagnosis of acute community-acquired pneumonia suggested by the presence of a cough, dirty sputum, chest pain and / or dyspnea (at least two criteria required), associated with the presence of a radiological or CT infiltrate initially
* Patient for whom it is not envisaged, a priori, to limit treatment within 5 days following inclusion, for ethical reasons, due to age and advanced comorbidities, and / or a level of severity beyond all therapeutic possibilities.
* Diagnosis of pneumonia done within 48 hours after admission to the hospital
* Participant admitted to the hospital for less than 8 days

"Control" group:

* Admission to the Intensive Care Units of the University Hospital of Tours or Limoges University Hospital
* Use of invasive mechanical ventilation for less than 48 hours
* Predictable duration of invasive mechanical ventilation> 48h
* Participant admitted to the hospital for less than 8 days
* Absence of pneumonia criteria (according to the criteria defined for the "Pneumonia" participant group)
* Absence shock (defined by the need for vasopressor despite volume expansion ≥30mL/kg, associated with a blood lactate level ≥ 2mmol / L
* Patient for whom it is not envisaged, a priori, to limit treatment within 5 days following inclusion, for ethical reasons, due to age and advanced comorbidities, and / or a level of severity beyond all therapeutic possibilities.

Exclusion Criteria:

* Participant under protection
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants admitted to the Intensive Care Unit of the University Hospital of Tours or University Hospital of Limoges (France) with an initial diagnosis of Community Acquired Pneumonia, or participants admitted without diagnosis of pneumonia or shock and for whom invasive mechanical ventilation is required.
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Blood level of Non-Conventional T Lymphocytes (expressed as % CD3+ lymphocytes) | 8 Months
Airway level of Non-Conventional T Lymphocytes (expressed as % CD3+ lymphocytes) | 8 Months
Blood level of inflammatory cytokines | 8 months
Airway level of inflammatory cytokines | 8 months

SECONDARY OUTCOMES:
Blood level of Conventional T Lymphocytes (expressed as % CD3+ lymphocytes) | 8 months
Airway level of Conventional T Lymphocytes (expressed as % CD3+ lymphocytes) | 8 months
Metabolic signature of non-conventional T lymphocytes | 8 months
Transcriptomic signature of non-conventional T lymphocytes | 8 Months
Blood level of Innate Cells (expressed as % CD45+ lymphocytes) | 8 months
AIrway level of Innate Cells (expressed as % CD45+ lymphocytes) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Youenn JOUAN, MD-PHD, Study Director — University of TOURS-INSERM U1100
Locations (3):
- France (3):
  - University Hospitakl of TOURS Département of Pneumonia, Tours
  - University Hospital -Bretonneau - Intensive Care, Tours
  - University Hospital of Tours; INSERM CIC 1415, Tours

IPD SHARING:
Plan to Share IPD: Undecided